CLINICAL TRIAL: NCT01273337
Title: A Phase 2 Randomized, Controlled Study With a Phase 1 Safety Cohort Testing ALD-401 Derived From Autologous Bone Marrow Delivered Via Intracarotid Infusion in Subjects With Ischemic Stroke With Blinded Assessments
Brief Title: Study of ALD-401 Via Intracarotid Infusion in Ischemic Stroke Subjects
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Aldagen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IS-001
Record Dates: First submitted 2011-01-06; First posted 2011-01-10 (Estimated); Last update posted 2014-01-16 (Estimated); Status verified 2014-01

CONDITIONS: Stroke; Ischemic Stroke; Stroke in Middle Cerebral Artery (MCA)
Keywords: Stroke; Ischemia; Ischemic Stroke; Middle Cerebral Artery; MCA; Stem Cells; Stem Cell; Autologous Bone Marrow; Ipsilateral MCA
MeSH Terms: conditions — Stroke; Ischemic Stroke; Ischemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ALD-401 (Experimental): ALD-401 is derived from Autologous Bone Marrow of the Stroke Subject
  Interventions: Biological: ALD-401
- Sham Comparitor (Sham Comparator): Sham Bone Marrow harvest and sham dosing procedure.
  Interventions: Procedure: Sham Procedure

INTERVENTIONS:
Biological: ALD-401 — 3 mL ALDHbr cells isolated from autologous bone marrow given as a one-time infusion via intracarotid infusion.
  Other Names: ALDHbr cells; ALDH Bright cells
  Arms: ALD-401
Procedure: Sham Procedure — Sham bone marrow harvest and sham product infusion procedures.
  Arms: Sham Comparitor

SUMMARY:
The purpose of this study is to demonstrate the safety of the delivery of ALD-401 by intracarotid infusion and to assess efficacy of treatment in subjects who have had unilateral, predominately cortical, ischemic strokes in the middle cerebral artery (MCA). ALD-401 is made from the stroke patient's bone marrow and infused 13-19 days after the stroke.

DETAILED DESCRIPTION:
This is a randomized, sham-controlled, multi-center, parallel-group, study in male and female subjects, designed to determine the safety and efficacy of ALD-401 in treating primary ischemic stroke. Approximately 100 subjects will be randomized 3:2 within a site to the treatment or sham control arm. Subjects experiencing an ischemic stroke will undergo either a bone marrow or a sham harvest on days 11-17 and be dosed with ALD-401 or a sham procedure 13-19 days after the primary event. Bone marrow cells are processed, sorted and formulated into a 3 mL suspension of ALD-401. Two days after harvest, subjects in the ALD-401 group will have their processed bone marrow cells (ALD-401) injected via intracarotid/MCA infusion, while control subjects have a sham infusion. All subjects will be followed for 12 months to monitor safety and to assess mental and physical function.

This study seeks to demonstrate safety of ALD-401 derived from autologous bone marrow and given via intracarotid delivery in a therapeutic window of 13-19 days post primary stroke event. This dosing window was selected to allow post-stroke inflammatory response to recede and therefore minimize the impact of resident inflammatory cells on the administration of ALD-401. This dosing window was consistent with information derived from pre-clinical models. Intracarotid/MCA delivery may offer minimal loss or dilution of therapeutic cells prior to localization in and around the ischemic area of the brain. ALD-401 will be manufactured from the patient's own bone marrow harvested 11-17 days after the primary stroke event.

ELIGIBILITY:
Inclusion Criteria:

1. Is age 30 to 83 years,
2. Has recent acute ischemic stroke in the middle cerebral artery (MCA) distribution confirmed by MRI or CT scan, with known onset time (within 24 hr),
3. Has persistent neurological deficit (NIHSS ≤22), mRS ≥ 3 at randomization,
4. Is able to provide bone marrow sample from anterior or posterior iliac crest at the time required by targeted infusion date,
5. Is able to return for dosing two days post bone marrow harvest (day 13-19 post stroke) and remain overnight for observation,
6. Is able to undergo (no contraindications) catheterization for localizing arteriograms for intracarotid/MCA delivery,
7. Has patency of the carotid artery on the affected side demonstrated at screening and prior to infusion; and flow is established in the proximal branches (M1 and M2) of the affected carotid if the stroke is cortical. Occlusion of either the M1 or M2 can be included in the study if imaging prior to harvest demonstrates flow through collateral circulation to the area of the infarct. If the infarction is lacunar, the proximal MCA must be patent,
8. Subjects who received tPA or underwent mechanical reperfusion may be included in the study as long as flow is established either in the proximal branches (M1 and M2) of the affected carotid or in the collateral circulation to the area of the infarct,
9. Has a general state that is compatible with a program of functional rehabilitation, and is receiving standard of care as determined by the investigator,
10. Is able to provide consent to study or informed consent is obtained from the subject's next of kin or legal representative,
11. Females must be postmenopausal, surgically sterilized, or practicing a suitable method of birth control so that, in the opinion of the investigator, they will not become pregnant during the course of the study,
12. Is a good candidate for the trial, in the opinion of the investigator.

Exclusion Criteria:

1. Medical Conditions:

   * Has a medical history of neurological or orthopedic pathology with deficit as a consequence that results in a modified Rankin Scale score >1 before stroke) or has a cognitive deficit,
   * Has a severe, persistent neurological deficit (NIHSS >22), OR a change of ≥4 points in the NIHSS from screening (after 7 days) to randomization (3-4 days after screening),
   * Has any clinically significant hemorrhagic (HI1 or PH1 petechial hemorrhages are allowed), or traumatic lesion of the brain on MRI or CT,
   * Has stroke affecting the sub cortical area only,
   * Has >50% stenosis or ulcerated plaque in the carotid artery on the ipsilateral side and carotid endarterectomy or arterial stenting is recommended for treatment,
   * Has had a seizure in the past 6 months (including associated with stroke),
   * Has a serious psychiatric disease which could alter evaluation on functional or cognitive scales,
   * Has a serious neurologic disease (e.g., multiple sclerosis, ALS) which could alter evaluation on functional or cognitive scales,
   * Had a myocardial infarction in the past 3 months,
   * Has a mechanical heart valve,
   * Has a history of ischemic stroke in any distribution within one month of the date of onset of the qualifying stroke for inclusion into this study,
   * Has known hepatic failure (Child-Pugh score Class B or C),
   * Has an active systemic infection,
   * Has an active malignancy or diagnosis of malignancy within 5 years prior to the start of screening (excluding skin cancers other than melanoma) or any history of chemotherapy or radiation affecting the bone marrow,
   * Has a history of inflammatory or progressively fibrotic conditions (e.g., rheumatoid arthritis, systemic lupus erythematosis, vasculitic disorders, idiopathic pulmonary fibrosis, retroperitoneal fibrosis),
   * Has another comorbid disease, including cardiovascular disease, which would be expected to result in less than 6-months life expectancy,
   * Has any concurrent illness or condition that in the opinion of the investigator might interfere with treatment or evaluation of safety and/or efficacy,
   * Has current or recent history of alcohol or drug abuse, or stroke considered associated with drug abuse.
2. Laboratory Findings:

   * Hemoglobin <10 g/dl,
   * Uncorrected coagulopathy as defined as INR >1.4; PTT >35 sec,
   * Platelet counts of <100,000 or >700,000,
   * Any hemodynamic instability at the time of consent (e.g., requiring continuous fluid resuscitation or ionotropic support), or hypoxemia (oxygen saturation of < 90%) on supplemental oxygen more than FIO2 = 0.3,
   * Renal insufficiency (creatinine clearance of < 50 mL/min/m2).
   * Poorly controlled diabetes mellitus (HbA1c > 10%),
   * Hypertension with SBP ≥ 150 mmHg or DBP ≥ 95 mmHg despite adequate anti-hypertensive treatment (at any measurement within 3 days of randomization).
3. Concomitant or Prior Therapies:

   * Subjects receiving systemic anticoagulation with warfarin, heparin or heparin analogs (patients on antiplatelet agents, including aspirin, or on prophylactic anticoagulation may enroll at the investigator's and proceduralists' discretion) and if exclusion 2b is not met,
   * Subjects currently receiving immunosuppressant drugs (e.g., for treatment of organ transplants, psoriasis, Crohn's disease, alopecia areata),
   * Subjects currently receiving restricted concomitant medications,
   * Any previous or current treatment with angiogenic growth factors, cytokines, gene therapy or stem cell therapy,
   * Currently receiving anti-angiogenic drugs,
   * Subjects participating in another clinical trial of an investigational therapy (including placebo) within 30 days of the start of screening.
4. Other:

   * Pregnant or nursing women (women capable of childbearing must have a negative serum pregnancy test at screening),
   * Is unable to return for follow up visits for clinical evaluation, safety evaluation, laboratory studies, or MRI or CT evaluation,
   * Is unable to undergo MRI or CT,
   * Has allergies to local or general anesthetics, or contrast media.

Ages: 30 Years to 83 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2011-03; Primary Completion 2014-07 (Estimated); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
Safety of Delivery of ALD-401 | 1 year
  The safety of the delivery of ALD-401 will be assessed by the following:
  * Frequency and proportion of severe adverse events,
  * Physical and clinical laboratory testing,
  * Radiological worsening as detected by MRI (evidence of hemorrhage) with and without clinical symptoms,
  * MRI evidence of new heterotopias, tumors, or vascular malformations over 12 months
  * Increase of NIHSS by ≥ 4 pts within 24 h of injection,
  * Re-hospitalization,
  * Survival.

SECONDARY OUTCOMES:
Efficacy of recovery of Mental and Physical Function | 1 year
  Determine the efficacy of ALD-401 for recovery of mental and physical function three months after treatment as assessed by the:
  * Modified Rankin Scale (mRS)
  * NIH Stroke Scale (NIHSS)
  * Barthel Index (BI)
  * European Quality of Life (EQ-5D)

CONTACTS AND LOCATIONS:
Overall Officials: James M Hinson, MD, Study Director — Aldagen
Locations (9):
- United States (9):
  - Los Angeles Brain and Spine Institute, Los Angeles, California
  - University of Miami Hospital, Miami, Florida
  - Minneapolis Heart Institute, Minneapolis, Minnesota
  - Duke University Medical Center, Durham, North Carolina
  - Ohio Health Research Institute, Columbus, Ohio
  - University of Pittsburgh Medical Center Presbyterian Hospital, Pittsburgh, Pennsylvania
  - University Medical Center at Brackenridge, Austin, Texas
  - The University of Texas Medical School, Houston, Texas
  - Swedish Medical Center, Cherry Hill Campus, Seattle, Washington

REFERENCES:
- [Derived] Savitz SI, Yavagal D, Rappard G, Likosky W, Rutledge N, Graffagnino C, Alderazi Y, Elder JA, Chen PR, Budzik RF Jr, Tarrel R, Huang DY, Hinson JM Jr. A Phase 2 Randomized, Sham-Controlled Trial of Internal Carotid Artery Infusion of Autologous Bone Marrow-Derived ALD-401 Cells in Patients With Recent Stable Ischemic Stroke (RECOVER-Stroke). Circulation. 2019 Jan 8;139(2):192-205. doi: 10.1161/CIRCULATIONAHA.117.030659. PMID 30586746